CLINICAL TRIAL: NCT00765583
Title: A Randomized, Evaluator-Blind, Multi-Center, Comparison of the Efficacy and Persistence of Correction of Nasolabial Folds With Restylane® Using Two Different Re-Treatment Schedules
Brief Title: A Study to Determine How Long Restylane® Will Last After Initial Treatment With 2 Different Re-treatment Schedules.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medicis Aesthetics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: MA-04-003; MA-04-003
Record Dates: First submitted 2008-10-01; First posted 2008-10-03 (Estimated); Last update posted 2011-09-22 (Estimated); Status verified 2011-09

CONDITIONS: Rhytids
Keywords: Wrinkles (Nasolabial Folds)
MeSH Terms: interventions — Restylane

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- restylane (Experimental): Restylane arm with different re-treatment schedules
  Interventions: Drug: Restylane

INTERVENTIONS:
Drug: Restylane — Treatment of the nasolabial folds with Restylane at Day 0/Baseline, Month 4.5, Month 9 and Month 18.

SUMMARY:
A total of 75 subjects will be enrolled into a 36 month study. Subjects will be treated with Restylane® on both sides of the face (nasolabial folds) at the first visit, on one side of the face at month 4.5 and on the other side of the face at month 9. Both sides of the face will then be treated again at month 18. The subjects will evaluate themselves and will also be evaluated by the treating doctor and a blinded evaluator (a person that does not know when the different sides of the face are treated). Side effects and medications taken during the study will also be recorded.

DETAILED DESCRIPTION:
The study will employ a randomized, evaluator-blind design. One of the nasolabial folds will be randomly assigned to be corrected with Restylane and then re-treated at 4 ½ months. The opposite side will be treated with Restylane and not re-treated until 9 months. Both nasolabial folds will be re-treated at 18 months. Each subject will serve as their own control, allowing comparison of the outcome between the contralateral sides.

This is a multi-center U.S. trial with a planned enrollment of 75 subjects at three centers. The goal of the study is to enroll and complete follow-up for 60 evaluable subjects. In order to compensate for early discontinuations, a total of at least 75 subjects will be recruited and treated.

After giving written informed consent, potential study participants will undergo a screening evaluation and initial treatment (Visit 1). The two nasolabial folds will be randomized for treatment so that one side will be designated for re-treatment with Restylane at 4 ½ months; the other at 9 months. At month 18 (Visit 7) both nasolabial folds will be re-treated. Follow-up visits will be scheduled through 36 months after initial treatment or touch-up.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

* Males or non-pregnant, non-breast feeding females aged 18 years or older.
* Subjects seeking augmentation therapy for correction of bilateral nasolabial folds.
* Subjects with a score of 3 or 4 on the Severity Rating Scale.
* Subjects with the ability to understand and comply with the requirements of the trial.
* Subjects willing to abstain from exclusionary procedures (e.g., further augmentation therapy,laser or chemical resurfacing; Botox® injections below eye level; facelift)for the duration of the study.
* Subjects willing to give written informed consent to participate in the trial.
* Women of childbearing potential must be willing to use an acceptable form of birth control during the study period.

Exclusion Criteria:

* Active or chronic skin disease, inflammation or related conditions, such as infection, psoriasis and herpes zoster near or on the nasolabial folds.
* Patients that have undergone procedures based on active dermal response (e.g. laser and chemical peeling procedures), within 6 months prior to study entry.
* Use of any facial tissue augmenting therapy or aesthetic facial surgical therapy within nine (9)months prior to study entry, e.g. injection or other form of implantation of tissue augmenting substances, Botox injections below the level of the eye-brows, facelift.
* Concomitant anticoagulant therapy, antiplatelet therapy, or a history of bleeding disorders.
* Patients who have previously experienced unanticipated adverse reactions when treated with hyaluronic acid based products.
* Any condition which in the opinion of the investigator makes the patient unsuitable for inclusion (e.g., patients not likely to avoid other treatments, patients not likely to stay in the study for six months, or patients anticipated to be unreliable).
* Subjects with cancerous or pre-cancerous lesions in the area to be treated.
* Use of any investigational drugs or devices within 30 days prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2005-11; Primary Completion 2008-12 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Blinded Evaluator Wrinkle Severity Rating Scale (WSRS) scores at month 18. | 18 months

SECONDARY OUTCOMES:
Subject and Blinded Evaluator WSRS scores at all other time points and Treating Investigator and Subject Global Aesthetic Improvement Scores (GAIS) at all time points. | Through end of study

CONTACTS AND LOCATIONS:
Overall Officials: Fredric Brandt, MD, Principal Investigator — Dermatology Research Institute, LLC; Steven Dayan, MD, Principal Investigator — Steven Dayan, MD; Rhoda narins, MD, Principal Investigator — Rhoda narins, MD
Locations (3):
- United States (3):
  - Dermatology Research Institute, LLC, Coral Gables, Florida
  - Dayan Facial Plastic Surgery Institute, Chicago, Illinois
  - Rhoda Narins, MD, White Plains, New York